CLINICAL TRIAL: NCT06060067
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Investigate the Safety and Immunogenicity of a Dengue Tetravalent Vaccine (Live, Attenuated) (TDV) Administered Subcutaneously to Healthy Subjects Aged 4 to 60 Years in India
Brief Title: A Study of Dengue Vaccine in Healthy Children, Teenagers and Adults in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DEN-302; 2023-000134-15 (EudraCT Number)
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: ≥18 to ≤60 Age Group: TDV (Experimental)
  Interventions: Biological: TDV
- Cohort 1: ≥18 to ≤60 Age Group: Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Cohort 2: ≥4 to <18 Age Group: TDV (Experimental)
  Interventions: Biological: TDV
- Cohort 2: ≥4 to <18 Age Group: Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TDV — TDV SC injection on Day 1 and Day 90 of the study
  Other Names: TAK-003
  Arms: Cohort 1: ≥18 to ≤60 Age Group: TDV; Cohort 2: ≥4 to <18 Age Group: TDV
Biological: Placebo — Normal Saline (0.9% NaCl) SC injection on Day 1 and Day 90 of the study
  Arms: Cohort 1: ≥18 to ≤60 Age Group: Placebo; Cohort 2: ≥4 to <18 Age Group: Placebo

SUMMARY:
The main aims of the study are to learn about side effects and a participant's immune response to Takeda's Dengue Vaccine when given twice within 3 months.

Participants will receive 2 doses of their randomized treatment (vaccine or placebo). Children, teenagers and adults will receive one dose of either the vaccine or placebo on Day 1 and the second dose of either the vaccine or placebo 3 months later. Up to 4 blood samples will be taken throughout the study.

During the study, participants will visit their study clinic 6 times.

DETAILED DESCRIPTION:
The vaccine being tested in this study is called TDV (Live, Attenuated). TDV is being tested to prevent dengue. This study will assess the safety and immunogenicity of TDV in healthy participants.

The study will enroll approximately 480 patients. Participants will be randomly assigned (by chance, like flipping a coin) to receive either TDV or placebo- which will remain undisclosed to the participant, and investigator during the study:

* Cohort 1, ≥18 to ≤60 Age Group: TDV
* Cohort 1, ≥18 to ≤60 Age Group: Placebo
* Cohort 2, ≥4 to <18 Age Group: TDV
* Cohort 2, ≥4 to <18 Age Group: Placebo

This multi-center trial will be conducted in India. The overall duration of the study is approximately 9 months.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants who can comply with trial procedures and are available for the duration of follow-up.

Key Exclusion Criteria:

At screening and at vaccination:

1. A body mass index (BMI) ≥35 kg/m^2.
2. Intent to participate in another clinical trial at any time during the conduct of this trial.
3. Plans to receive any of the following:

   1. A licensed vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to TDV or placebo administration.
   2. A coronavirus vaccine within 14 days prior to TDV or placebo administration.
   3. A vaccine authorized for emergency use within 28 days of TDV or placebo administration.
4. Known substance or alcohol abuse within the past 2 years that may interfere with his/her ability to comply with requirements for trial participation.
5. Receipt of previous vaccination against dengue virus.
6. Previous participation in any clinical trial of a dengue candidate vaccine.

At Vaccination:

1. Participants with febrile illness or moderate or severe acute illness, or infection, at the time of random assignment.
2. Participants medicated with antipyretic and/or analgesic medication(s) within 24 hours prior to TDV or placebo administration.

NOTE: Other protocol defined Inclusion/exclusion criteria may apply.

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 480 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local (Injection Site) Adverse Events (AEs) by Severity Within 7 Days Post Vaccination at Day 1 | Within 7 days postvaccination at Day 1
  Solicited local AEs at injection site are defined as injection site pain, injection site erythema, and injection site swelling. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Number of Participants with Solicited Local Injection Site AEs, by Severity Within 7 Days Post Vaccination at Day 90 | Within 7 days postvaccination at Day 90
  Solicited local AEs at injection site are defined as injection site pain, injection site erythema, and injection site swelling. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Number of Participants with Solicited Systemic AEs by Severity Within 14 Days Post Vaccination at Day 1 | Within 14 days postvaccination at Day 1
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. Solicited systemic AEs assessments for children <6 years old include: drowsiness, irritability/fussiness, loss of appetite and fever, and those for children ≥ 6 years old/adolescent/adult include: headache, asthenia, malaise, myalgia and fever. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Number of Participants with Solicited Systemic AEs, by Severity Within 14 Days Post Vaccination at Day 90 | Within 14 days postvaccination at Day 90
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. Solicited systemic AEs assessments for children <6 years old include: drowsiness, irritability/fussiness, loss of appetite and fever, and those for children ≥ 6 years old/adolescent/adult include: headache, asthenia, malaise, myalgia and fever. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Any Unsolicited AEs Within 28 Days Post Vaccination at Day 1 | Within 28 days postvaccination at Day 1
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Percentage of Participants with Any Unsolicited AEs Within 28 Days Post Vaccination at Day 90 | Within 28 days postvaccination at Day 90
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Percentage of Participants with an AE Leading to Participant Withdrawal from Trial | From first vaccination on Day 1 through the end of trial (up to Day 270)
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Percentage of Participants with an AE Leading to TDV or Placebo Discontinuation. | From first vaccination on Day 1 through the end of trial (up to Day 270)
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Percentage of Participants with a Medically-attended AE (MAAE) | From first vaccination on Day 1 through the end of trial (up to Day 270)
  MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria.
Percentage of Participants with a Serious Adverse Event (SAE) | From first vaccination on Day 1 through the end of trial (up to Day 270)
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An SAE is defined as any untoward medical occurrence that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/ incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, is an important medical event.
Geometric Mean Titers (GMTs) of Neutralizing Antibodies by Microneutralization Test for Each of the 4 Dengue Virus Serotypes | Day 120 (Month 6)
  GMTs of neutralizing antibodies will be measured by microneutralization test 50% [MNT50] for each of the 4 Dengue Serotypes for all participants. The 4 dengue virus serotypes are dengue virus (DENV)-1, DENV-2, DENV-3 and DENV-4.

SECONDARY OUTCOMES:
Geometric Mean Titers by Microneutralization Test for Each of the 4 Dengue Virus Serotypes | Day 1 and Day 270
  GMTs of neutralizing antibodies will be measured by MNT50 for each of the 4 Dengue Serotypes for all participants. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Percentage of Participants With Seroconversion for Each of the 4 Dengue Virus Serotypes | Day 1, Day 120 and Day 270
  Seroconversion rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositive is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Percentage of Participants With Seroconversion for Multiple (2, 3, or 4) Dengue Virus Serotypes | Day 1, Day 120 and Day 270
  Seroconversion rate, defined as the percentage of participants seropositive, is derived from the titers of dengue-neutralizing antibodies. Seropositive is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- India (10):
  - BGS Global Institute of Medical Sciences (BGS-GIMS) #67, BGS Health & Education City, Uttarahalli Main Road, Kengeri, Bangalore, Karnataka
  - Chettinad Academy of Research and Education, Chettinad Health City, SH,49A, Dist. Kelambakkam, Pudupākkam, Tamil Nadu
  - Preventive and Therapeutic Clinical Trial Unit (PTCTU), Dept. of Community Medicine, Institute of Medical Science and SUM Hospital, K-8, Kalinga Nagar, Bhubaneshwar
  - SRM Medical College Hospital & Research Centre, SRM Nagar, Potheri, Kattankulathur
  - IPGME&R and SSKM Hospital, 244 AJC Bose Road, Kolkata
  - King George's Medical University, Department of Medicine, Chowk, Lucknow
  - Suyog Hospital, 2nd Floor, B-Wing, Krushi Utpanna Bazar, Samiti Sankul, Dindori Rd, Panchavati, Nashik
  - Maulana Azad Medical College & Associated Lok Nayak, Govind Ballabh Pant Hospitals and Guru Nanak Eye Center, New Delhi
  - KEM Hospital Research Centre, Sandar Moodliar Road, Rasta Peth, Pune
  - King George Hospital, Visakhapatnam

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/6d91b0e82e6c410b?idFilter=%5B%22DEN-302%22%5D